CLINICAL TRIAL: NCT04264585
Title: Examining Motivational Interviewing and Booster Sessions in Internet-delivered Cognitive Behaviour Therapy for Post-secondary Students: An Implementation Trial
Brief Title: Internet-delivered Cognitive Behaviour Therapy (ICBT) for Post-secondary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2019-205
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; post-secondary students; internet-delivered cognitive behaviour therapy; randomized controlled trial; patient-centred; therapist-assistance
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard ICBT (Experimental): Clients assigned to the Standard ICBT condition will receive the standard version of the ICBT course, which consists of four lessons spread across the span of five weeks. Clients will receive five weeks of therapist support.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- ICBT with Motivational Interviewing (Experimental): Clients assigned to the ICBT with Motivational Interviewing condition will receive the Planning for Change lesson before Lesson 1 of the UniWellbeing Course.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy; Behavioral: Motivational Interviewing
- ICBT with Booster (Experimental): Clients assigned to the ICBT with Booster condition will receive access to a booster session one month after the end of the ICBT course.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy; Behavioral: Booster Session
- ICBT with Motivational Interviewing and Booster (Experimental): Clients assigned to the ICBT with Motivational Interviewing and Booster condition will receive access to both the Motivational Interviewing content (before Lesson 1 of the UniWellbeing Course) and the booster session (one month after ICBT course).
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy; Behavioral: Motivational Interviewing; Behavioral: Booster Session

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behaviour therapy — All clients will receive the same materials, namely the UniWellbeing Course, which was developed at Macquarie University, Australia. The UniWellbeing Course is a transdiagnostic intervention targeting symptoms of depression and anxiety, that has been tailored for use in post-secondary students. It comprises 4 online lessons that provide psychoeducation about: symptom identification and the cognitive behavioural model; thought monitoring and challenging; de-arousal strategies and pleasant activity scheduling; graduated exposure; and relapse prevention. Seven supplementary lessons can also be accessed at any time (e.g., sleep, communication). Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills) with 4 lesson summaries and homework assignments that facilitate skill acquisition. Therapists will spend ~15 mins. per week/per client.
Behavioral: Motivational Interviewing — Clients assigned to the ICBT with Motivational Interviewing condition will receive access to the Planning for Change lesson before accessing Lesson 1. They will be presented with five interactive online exercises based on motivational interviewing principles (i.e. values clarification, importance ruler, looking back, confidence ruler, and looking forward). As clients complete the exercises, they are prompted to answer open-ended questions and are provided with written feedback.
  Arms: ICBT with Motivational Interviewing; ICBT with Motivational Interviewing and Booster
Behavioral: Booster Session — Clients assigned to the ICBT with Booster condition will receive access to a booster session one month after the end of the ICBT course. The booster session will include information about maintaining motivation, a review of the ICBT course content and skills, and information about structured problem solving. Clients will also have access to a Do-It-Yourself guide that summarizes the information in the booster session and includes worksheets for clients to practice the problem-solving skills described in the booster.
  This booster session will be self-guided (ie. no therapist support is offered).
  Arms: ICBT with Booster; ICBT with Motivational Interviewing and Booster

SUMMARY:
Post-secondary students are at an elevated risk for anxiety and depression, with approximately one in three students experiencing clinical levels of symptoms at some point during their academic career. Despite the high prevalence of these mental health concerns, many students do not receive adequate treatment. Internet-delivered cognitive behaviour therapy (ICBT) is an alternative to face-to-face service that is effective for improving symptoms of anxiety and depression in general adult populations. Recently, there has been increasing interest in the use of ICBT in post-secondary populations, however high drop-out rates and small effect sizes suggest that current ICBT programs are not fully meeting students' specific needs. Additional research is necessary to ensure that ICBT is delivered to students in a manner that is both acceptable and effective.

The proposed study will be an implementation trial to examine whether the efficacy of an ICBT course for post-secondary students is improved by offering a motivational interviewing component at pre-treatment and a booster session 1-month after completing treatment. Follow-up assessment will be conducted as 3-month post-treatment. Primary outcomes are anxiety, depression, and academic functioning. Implementation outcomes will include measures of the acceptability, adoption, and fidelity (assessed by number of modules completed) of the ICBT course.

DETAILED DESCRIPTION:
The aims of the study will be to: assess the efficacy of the UniWellbeing Course in reducing symptoms of anxiety and depression and increasing adjustment to academic and social responsibilities; to assess the impact of a pre-treatment motivational interviewing component on attrition, engagement, and outcomes (depression, anxiety, and academic functioning); to assess the impact of a booster session on anxiety, depression, and academic and social adjustment at three-month follow-up; and to assess the combined effect of including both a motivational interviewing component and booster session on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* registered as a student at a post-secondary institution in Saskatchewan; over the age of 18;endorse symptoms of depression and/or anxiety; be able to access computers and the Internet and be comfortable using them; and willing to provide a physician as an emergency contact

Exclusion Criteria:

* high risk of suicide or hospitalization for mental health in previous 12 months
* unmanaged alcohol or drug use problems
* severe psychiatric illness that is not managed (e.g. psychosis or mania)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline (screening), weeks 1-6, 9, and 17
  Change in depression symptoms. 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (screening), weeks 1-6, 9, and 17
  Change in anxiety symptoms. 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Sheehan Disability Scale (SDS) | Baseline (screening), week 6, 9, and 17
  Change in disability. Three items are summed into a total score ranging from 0 to 30, with higher scores indicating higher levels of disability.
Alcohol Use Disorders Identification Test (AUDIT) | Baseline (screening), week 6, and week 9
  A 10-item screening tool to assess alcohol consumption. Items 1 to 8 are scored on a scale ranging from 0 to 4. Items 9 and 10 are scored on a three-point scale (0, 2, or 4). Scores from 10 items are summed with possible scores ranging from 0 to 40 and higher scores indicating a higher likelihood of problematic alcohol consumption.
Drug Use Disorders Identification Test (DUDIT) | Baseline (screening), week 6, and week 9
  An 11-item screening tool to assess problematic drug use. Items 1 to 9 are scored on a scale ranging from 0 to 4. Items 10 and 11 are scored as a 0, 2, or 4. Total scores for the DUDIT range from 0 to 44 with higher scores suggesting problematic drug use.
Academic functioning | Baseline (screening), weeks 1-6, 9, and 17
  Self-report measure of self-efficacy for academic functioning/skills. Items are scored from 0-10, with higher scores indicating higher levels of perceived self-efficacy.
Treatment credibility. | Baseline (screening), week 6
  Measured by Treatment Credibility Questionnaire (TCQ) which contains 4 items. The first three items range from 0-9 with higher scores indicating better outcome, and the fourth item ranges from 0-100%, with higher scores indicating greater improvement in functioning.
Treatment satisfaction | Week 6
  Measured by Internet-CBT Treatment Satisfaction Measure. Measure includes 19 questions assessing satisfaction with various aspects of Internet-CBT and also negative effects of treatment
Change Questionnaire | Pre-treatment
  The CQ is a self-report measure that focuses on three factors of change: importance, ability, and commitment. For the purpose of this study, the desired change will be to "reduce the anxiety and/or depression I experience". For each of the three factors, participants are asked to rate on a scale of 0 ("Definitely not") to 10 ("Definitely") how motivated they are to make the change. Total scores on the questionnaire can range from 0 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Peynenburg, MA, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit University of Regina, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Peynenburg V, Hadjistavropoulos H, Thiessen D, Titov N, Dear B. Internet-Delivered Cognitive Behavioral Therapy for Postsecondary Students: Randomized Factorial Trial for Examining Motivational Interviewing and Booster Lessons. J Med Internet Res. 2022 Sep 7;24(9):e40637. doi: 10.2196/40637. PMID 36069785